CLINICAL TRIAL: NCT05092750
Title: Magnetic Particle-ICG Lymph Node Mapping in Colorectal Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: 0 accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-0479
Record Dates: First submitted 2021-09-21; First posted 2021-10-26 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FerroTraceTM (magnetic tracer) (Experimental): a special type of fluorescent dye called indocyanine green (ICG) during surgery can help surgeons find the lymph nodes that the cancer is most likely to have spread to in colorectal cancer patients.
  Interventions: Device: FerroTraceTM; Drug: indocyanine green (ICG)

INTERVENTIONS:
Device: FerroTraceTM — A magnetic
Drug: indocyanine green (ICG) — Given by SC injection

SUMMARY:
Study to determine the feasibility of Sentinel Lymph Node (SLN) mapping using novel magnetic tracers (FerroTrace) and indocyanine green (ICG) for colorectal cancer; and to evaluate safety by assessing short term toxicity associated with colonoscopic peritumoral injection of novel magnetic nanoparticles (FerroTrace) and ICG for colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY:

1. To determine the feasibility of Sentinel Lymph Node (SLN) mapping using novel magnetic tracers (FerroTrace) and indocyanine green (ICG) for colorectal cancer.
2. To evaluate safety by assessing short term toxicity associated with colonoscopic peritumoral injection of novel magnetic nanoparticles (FerroTrace) and ICG for colorectal cancer.

SECONDARY:

1. To determine the additional positive diagnostic value of adding sentinel lymph node mapping to lymphadenectomy by assessing the SLNs with detailed immunochemistry versus the normal H&E staining pathology tests.

PRIMARY END POINTS:

1. Feasibility: Number of registered patients who complete all study procedures with at least one sentinel node identified.
2. Safety: Rate of any grade III or greater toxicity attributable to FerroTrace injection, evaluated using the Common Terminology Criteria for Adverse Events (CTCAE) v. 5.0. Adverse events according to general peri-operative complications.

SECONDARY ENDPOINTS:

1. The identification rate and number of FerroTrace-positive lymph nodes for each patient.
2. Incidence of pathological upstaging of LN metastasis status by the addition of (non-routine) serial H&E and immunohistochemistry in the pathological assessment of identified FerroTrace-positive lymph nodes.

ELIGIBILITY:
Inclusion criteria:

* Age 18 or older
* Willing to provide informed consent
* Biopsy proven colon or rectal cancer
* No distant metastases

Exclusion criteria:

* Serious medical comorbidities or other contraindications to surgery +/- adjuvant therapy as determined by the treatment team
* Previous pelvic radiotherapy or radiotherapy planned prior to surgery
* Allergy or intolerance to iron oxide compounds
* Iron overload disorder
* Allergy or intolerance to iodides
* Pregnant or lactating women*

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2023-08-29 (Actual); Study Completion 2023-08-29 (Actual)

PRIMARY OUTCOMES:
To assess the feasibility how the Sentinel Lymph Node (SLN) mapping by using novel magnetic tracers (FerroTrace) and using the indocyanine green (ICG) for colorectal cancer. | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: George Chang, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org